CLINICAL TRIAL: NCT00671827
Title: Prospective Evaluation of Robot-Assisted Surgery in Gynecologic Oncology
Brief Title: Evaluation of Robot-Assisted Surgery in Gynecologic Oncology
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0122
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer; Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Uterine Cancer; Vaginal Cancer; Vulvar Cancer; Questionnaire; Survey; Robot-Assisted Surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robotic Gynecologic Surgery: Patients who have undergone or will undergo a robotic-assisted gynecologic procedure.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires each taking less than 10 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this observational study is to collect information about the length of surgery, the procedures performed during surgery, and any possible side effects of robot-assisted gynecologic cancer surgeries. The researchers also want to learn if patients who have robot-assisted surgeries have fewer complications during recovery.

DETAILED DESCRIPTION:
Information Collection:

If you agree to take part in this study, the following information will be collected from your medical record after surgery:

* The reason you had or are scheduled to have robot-assisted surgery.
* How long the surgery took to complete.
* What procedures were performed during the surgery.
* If cancer was or was not found in the tissue that was removed.
* How long you were in the hospital.
* What complications, if any, happened that are related to the surgery.

Follow-Up Questionnaires:

Depending on when you enroll in the study, you may be asked to complete a short questionnaire 3 different times, each questionnaire will take less than 10 minutes to complete. If you had surgery for cervical cancer, you will complete the questionnaire 2 weeks after surgery. All patients will complete the questionnaires 4-6 weeks after surgery, and again 3-6 months later.

If you have your follow up care with a doctor outside of MD Anderson, you will be called to complete the questionnaires over the phone. Each phone call should last about 10 minutes This questionnaire and/or phone calls will ask questions about any side effects you have experienced that you think may be related to the surgery.

Length of Study:

After the last questionnaire is completed, your participation in the study is over.

This is an investigational study.

Up to 1,000 patients will take part in this study at MD Anderson Cancer Center and Banner MD Anderson Arizona.

ELIGIBILITY:
Inclusion Criteria:

1) All women who have undergone or will undergo a robotic-assisted gynecologic procedure at MD Anderson Cancer Center and MD Anderson Banner - Arizona are eligible for inclusion in this study. They should be able to speak either English or Spanish.

Exclusion Criteria:

1) None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who have undergone or will undergo a robotic-assisted gynecologic procedure at M. D. Anderson Cancer Center and St. Luke's Episcopal Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2008-04-29 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Data Collection of Surgical Times, Procedures Performed, Intra-operative + Postoperative Complications of Robot-assisted Gynecologic Oncology Cases | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Soliman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - MD Anderson Banner Arizona, Gilbert, Arizona
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org